CLINICAL TRIAL: NCT02583269
Title: Phase I Study of Muscadine Grape Extract (MGE) in Advanced Malignancy
Brief Title: Muscadine Grape Skin Extract in Treating Patients With Malignancy That Is Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00035394; NCI-2015-01710 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01815 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-22 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm; Unresectable Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1 (muscadine grape skin extract) 1 pill 2 times a day (Experimental): Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Diagnostic Test: Laboratory Biomarker Analysis; Drug: Muscadine Grape Skin Extract; Procedure: Quality-of-Life Assessment
- Arm 2 (muscadine grape skin extract) 2 pills 2 times a day (Experimental): Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Diagnostic Test: Laboratory Biomarker Analysis; Drug: Muscadine Grape Skin Extract; Procedure: Quality-of-Life Assessment
- Arm 3 (muscadine grape skin extract) 3 pills 2 times a day (Experimental): Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Diagnostic Test: Laboratory Biomarker Analysis; Drug: Muscadine Grape Skin Extract; Procedure: Quality-of-Life Assessment
- Arm 4 (muscadine grape skin extract) 4 pills 2 times a day (Experimental): Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Diagnostic Test: Laboratory Biomarker Analysis; Drug: Muscadine Grape Skin Extract; Procedure: Quality-of-Life Assessment
- Arm 5 muscadine grape skin extract) 5 pills 2 times a day (Experimental): Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Diagnostic Test: Laboratory Biomarker Analysis; Drug: Muscadine Grape Skin Extract; Procedure: Quality-of-Life Assessment

INTERVENTIONS:
Diagnostic Test: Laboratory Biomarker Analysis — Correlative studies
Drug: Muscadine Grape Skin Extract — Given PO
  Other Names: MSKE
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I trial studies the side effects and the best dose of muscadine grape skin extract (MGE) in treating patients with malignancy (tumor or cancer) that has spread to other parts of the body or cannot be removed by surgery. MGE is a nutritional supplement containing an extract of the skin of muscadine grape that has shown anti-cancer activity in laboratory studies and may be able to fight or kill malignant cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and maximum tolerated dose (MTD) of MGE (muscadine grape skin extract) after 4 weeks of administration for patients with metastatic cancer.

Secondary Objectives:

I. To monitor adverse events/toxicity every 4 weeks while on treatment. II. To evaluate change in phenolic levels (total and component, blood and urine) from baseline to 4 and 8 weeks.

III. To evaluate change in serum cytokines and growth factors from baseline to 4 and 8 weeks on MGE.

IV. To observe the response rate of MGE in patients with metastatic cancer. V. To assess overall and progression-free survival in patients with metastatic cancer receiving MGE.

VI. To assess global quality of life (Functional Assessment of Cancer Therapy-General [FACT-G] and fatigue (Patient Reported Outcomes Measurement Information System [PROMIS]-fatigue Short Form [SF]) in cancer patients taking MGE.

VII. To assess adherence to MGE treatment.

OUTLINE: This is a dose-escalation study.

Patients receive muscadine grape skin extract orally (PO) twice daily (BID). Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and have failed standard therapies
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1000/mcL
* Platelets >= 50,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit or normal
* Creatinine clearance >= 40 mL/min
* Stable supplement usage for > 2 weeks prior to starting and agrees not to change while on this study
* Life expectancy > 3 months

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational cancer-directed agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MGE
* Patients unable to take oral medications or those with history of malabsorption due to bowel resection
* Patients with uncontrolled diarrhea or persistent nausea/vomiting requiring daily antiemetic therapy for symptom management
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued
* Patients with primary brain tumors are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Bitting RL, Tooze JA, Isom S, Petty WJ, Grant SC, Desnoyers RJ, Thomas A, Thomas CY, Alistar AT, Golden SL, Pleasant K, Chappell MC, Tallant EA, Gallagher PE, Klepin HD. Phase I Study of Muscadine Grape Extract for Patients With Advanced Cancer. Am J Clin Oncol. 2021 Jun 1;44(6):239-246. doi: 10.1097/COC.0000000000000814. PMID 33867481

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Muscadine Grape Skin Extract) 1 Pill 2 Times Per Day; Arm 2 (Muscadine Grape Skin Extract) 2 Pills 2 Times a Day; Arm 3 (Muscadine Grape Skin Extract) 3 Pills 2 Times a Day; Arm 4 (Muscadline Grape Skin Extract) 4 Pills 2 Times a Day; Arm 5 (Muscadine Grape Skin Extract) 5 Pills 2 Times a Day: Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Muscadine Grape Skin Extract: Given PO
  Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Arm 1 (Muscadine Grape Skin Extract) 1 Pill 2 Times Per Day | Arm 2 (Muscadine Grape Skin Extract) 2 Pills 2 Times a Day | Arm 3 (Muscadine Grape Skin Extract) 3 Pills 2 Times a Day | Arm 4 (Muscadline Grape Skin Extract) 4 Pills 2 Times a Day | Arm 5 (Muscadine Grape Skin Extract) 5 Pills 2 Times a Day
Started | 3 | 7 | 3 | 5 | 6
Completed | 2 | 7 | 3 | 5 | 6
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Patient hospitalized prior to start | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 (Muscadine Grape Skin Extract) 1 Pill Times a Day; Arm 2 (Muscadine Grape Skin Extract) 2 Pills Times a Day; Arm 3 (Muscadine Grape Skin Extract) 3 Pills Times a Day; Arm 4 (Muscadine Grape Skin Extract) 4 Pills Times a Day; Arm 5 (Muscadine Grape Skin Extract) 5 Pills Times a Day: Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Muscadine Grape Skin Extract: Given PO
  Quality-of-Life Assessment: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Muscadine Grape Skin Extract) 1 Pill Times a Day | Arm 2 (Muscadine Grape Skin Extract) 2 Pills Times a Day | Arm 3 (Muscadine Grape Skin Extract) 3 Pills Times a Day | Arm 4 (Muscadine Grape Skin Extract) 4 Pills Times a Day | Arm 5 (Muscadine Grape Skin Extract) 5 Pills Times a Day | Total
Number analyzed (Participants) | 3 | 7 | 3 | 5 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.3 (3.29) | 73.4 (13.56) | 62.6 (6.24) | 64 (7.13) | 70 (11.8) | 69.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 3 | 2 | 10
  Male | 3 | 4 | 1 | 2 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 7 | 3 | 5 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 2 | 7 | 3 | 5 | 6 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 3 | 5 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity
Description: Maximum tolerable dose of muscadine grape extract is defined as the dose level immediately below the dose level that induced a dose-limiting toxicity (DLT) in >= 2 patients, as assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0DLT will be assessed by severity of adverse events.
Time Frame: 29 days
Population: As pre-specified in the protocol, data collection and analysis for all arms will be combined. MTD was not determined, as there was not a dose level with ≥2 dose limiting toxicities (DLT). One DLT at dose level 2 and therefore 3 additional participants were enrolled. No subsequent DLTs and the study was stopped at dose level 5, per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Muscadine Grape Skin Extract) 1 Pill 2 Times Per Day | Arm 2 (Muscadine Grape Skin Extract) 2 Pills 2 Times a Day | Arm 3 (Muscadine Grape Skin Extract) 3 Pills 2 Times a Day | Arm 4 (Muscadline Grape Skin Extract) 4 Pills 2 Times a Day | Arm 5 (Muscadine Grape Skin Extract) 5 Pills 2 Times a Day
Number analyzed (Participants) | 3 | 7 | 3 | 5 | 6
Participants | 0 | 1 | 0 | 0 | 0

2. Secondary Outcome: Adherence to MGE Treatment, as Measured by Percent of Pills Taken at the End of Every 4 Week Period
Description: Pill count will be calculated from counting the number of pills returned as well as by summarizing the patient's pill diary. The percent of pills taken will be summarized by dose level using the median and 95% confidence interval. Investigators will summarize the percent of pills taken at the end of every 4 week period i using the formula: Percent of pills taken)i = (Dose Level ×7 ×4)i minus Pill Count divided by Dose Level ×7 ×4)i
Time Frame: Up to 1 year
Population: As pre-specified in the protocol, this study is not intended to be analyzed by arm for most analyses and data collection. Analysis for all arms will be combined for Adherence to EMG treatment.
Measure: Median (95% Confidence Interval); unit: percentage of pills
Groups:
- Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS: Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Muscadine Grape Skin Extract: Given PO
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 19
percentage of pills | 97.8 [95.8 to 99.4]

3. Secondary Outcome: Best Response
Description: Best response will be characterized using a frequency table. Evaluation of new or enlarging effusions to differentiate between Progressive Disease and Response/Stable Disease. Measurements will be obtained from usual care imaging and assessed by the principal investigators in confirmation with the physician of record. Clinical lesions will only be considered measurable when they are superficial and ≥10 mm in diameter as assessed using calipers. For the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.
Time Frame: At the end of treatment, up to 1 year
Population: As pre-specified in the protocol, this study is not intended to be analyzed by arm for most analyses and data collection. Analysis for all arms will be combined for Best Response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 16
Participants
  Stable Disease | 8
  Progressive Disease | 8

4. Secondary Outcome: Change in Total Phenolic Levels in Blood
Description: A mixed model analysis of variance (ANOVA) model will be fit with phenolic level as the outcome and time (baseline, 4, and 8 weeks) as a fixed effect and subject as a random effect. Contrasts will be used to estimate the changes from baseline to week 4 and week 8.
Time Frame: Baseline to up to 8 weeks
Population: As pre-specified in the protocol, this study is not intended to be analyzed by arm for most analyses and data collection. Analysis for all arms will be combined for change in total phenolic levels in blood.
Measure: Mean (Standard Error); unit: ug/ml
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 19
ug/ml
  Baseline | 2123.8 (69.1)
  Week 4 | 2049.3 (69.1)
  Week 8 | 2308.1 (71.7)

5. Secondary Outcome: Change in Total Phenolic Levels in Urine
Description: as for outcome 4
Time Frame: Baseline to up to 8 weeks
Population: Arms were combined for cytokine and phenolic analyses as pre-specified per protocol
Measure: Mean (Standard Error); unit: ug/ml
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 19
ug/ml
  Baseline | 1107.2 (142.4)
  Week 4 | 1024.5 (142.3)
  Week 8 | 1274.6 (150.7)

6. Secondary Outcome: Change in Quality of Life and Fatigue in Cancer Patients Taking MGE as Measured by FACT-G
Description: A mixed model ANOVA model will be fit with phenolic level as the outcome and time (baseline, every 4 weeks) as a fixed effect and subject as a random effect. Contrasts will be use to estimate changes from baseline to each follow-up time period. Score scales from 0 (not at all) to 4 (very much). Sum of scores range 0-28 for social, functional and physical well being and 0-24 for emotional well being and multiplied by 6. All four scores are totaled with a score range of 0-108. A mean of the combined group scores will be used. A higher score indicates a higher worse outcome of the illness on the participant.
Time Frame: Baseline to up to 1 year
Population: As pre-specified in the protocol, this study is not intended to be analyzed by arm for most analyses and data collection. Analysis for all arms will be combined for change in quality of life. All participants did not complete intervention for outcome measures are various time points (i.e., week 4 and week 8)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 21
score on a scale
  FACT-G Overall Score - at Baseline | 80.6 (3.9)
  Fact G - Overall Score - at Week 4: number analyzed (Participants) | 19
  Fact G - Overall Score - at Week 4 | 79.4 (3.9)
  Fact G - Overall Score - at Week 8: number analyzed (Participants) | 13
  Fact G - Overall Score - at Week 8 | 81.1 (4.0)
  Functional well being - at Baseline | 17.7 (1.6)
  Functional well being - at Week 4: number analyzed (Participants) | 19
  Functional well being - at Week 4 | 17.7 (1.6)
  Functional well being - at Week 8: number analyzed (Participants) | 13
  Functional well being - at Week 8 | 16.5 (1.7)
  Emotional Well being - at Baseline | 17.8 (0.9)
  Emotional well being - at Week 4: number analyzed (Participants) | 19
  Emotional well being - at Week 4 | 17.8 (0.9)
  Emotional well being - at Week 8: number analyzed (Participants) | 13
  Emotional well being - at Week 8 | 18.8 (1.0)
  Physical well being - at Baseline | 20.6 (1.5)
  Physical well being - at Week 4: number analyzed (Participants) | 19
  Physical well being - at Week 4 | 19.3 (1.5)
  Physical well being - at Week 8: number analyzed (Participants) | 13
  Physical well being - at Week 8 | 20.4 (1.6)
  Social well being - at Baseline | 24.5 (0.7)
  Social well being - at Week 4: number analyzed (Participants) | 19
  Social well being - at Week 4 | 24.9 (0.7)
  Social well being - at Week 8: number analyzed (Participants) | 13
  Social well being - at Week 8 | 25.4 (0.8)
Statistical Analysis 1: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Overall FACT G score p value baseline to week 8; Test type: Other; p = 0.76, ANOVA
Statistical Analysis 2: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Fact G functional well being p value baseline to week 8; Test type: Other; p = 0.25, ANOVA
Statistical Analysis 3: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; FACT G emotional well being p value baseline to week 8; Test type: Other; p = 0.18, ANOVA
Statistical Analysis 4: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Fact G physical well being p value baseline to week 8; Test type: Other; p = 0.87, ANOVA
Statistical Analysis 5: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Fact G social well being p value baseline to week 8; Test type: Other; p = 0.22, ANOVA

7. Secondary Outcome: Change in Systemic Cytokine Levels
Description: A mixed model ANOVA model will fit with the outcome of interest (cytokine or growth factor) as the outcome and time (baseline, 4, and 8 weeks) as a fixed effect and subject as a random effect. Contrasts will be used to estimate the changes from baseline to week 4 and week 8.
Time Frame: Baseline to up to 8 weeks
Population: Arms were combined for cytokine and phenolic analyses as pre-specified per protocol
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 19
pg/mL
  Baseline to Week 8 IL-1 alpha | NA (NA) — All values below lower limit of detection - could not be analyzed
  Baseline to 8 weeks IL-1 beta | NA (NA) — 70% of values below lower limit of detection - could not be analyzed
  Baseline to 8 weeks IL-6 | NA (NA) — 85% of values below lower limit of detection - could not be analyzed
  Baseline TNF alpha | 4.74 (0.39)
  Week 4 TNF alpha | 4.95 (0.39)
  Week 8 TNF alpha | 4.97 (0.41)
  Baseline IL-6R | 10905.9 (1013.7)
  Week 4 IL-6R | 11111.7 (993.7)
  Week 8 IL-6R | 12402.9 (1077.9)

8. Secondary Outcome: Incidence of Adverse Events (AEs), Assessed Using NCI CTCAE Version 4.0
Description: AEs/toxicity will be assessed at weeks 4, 8 and every 4 weeks thereafter if patients remain on treatment. Any expected toxicities, any laboratory based toxicities, and any grade 3 or higher gastrointestinal toxicities, and any grade 4 or higher toxicities will be summarized using frequency tables overall and by week.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Muscadine Grape Skin Extract) 1 Pill 2 Times Per Day | Arm 2 (Muscadine Grape Skin Extract) 2 Pills 2 Times a Day | Arm 3 (Muscadine Grape Skin Extract) 3 Pills 2 Times a Day | Arm 4 (Muscadline Grape Skin Extract) 4 Pills 2 Times a Day | Arm 5 (Muscadine Grape Skin Extract) 5 Pills 2 Times a Day
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 6
Participants | 3 | 3 | 2 | 2 | 5

9. Secondary Outcome: Overall Response Rate of MGE (Complete Response, Partial Response, and Stable Disease)
Description: Response will be characterized using a frequency table.
Time Frame: At 8 weeks
Population: As pre-specified in the protocol, data will be collected and analyzed for all arms combined. At 8 weeks, only 16 patients were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 16
Participants
  Stable Disease | 8
  Progressive Disease | 8

10. Secondary Outcome: Overall Survival (OS)
Description: OS will summarized using the Kaplan-Meier method. Median survival rates and associated 95% confidence intervals will be calculated.
Time Frame: Up to 4 years
Population: As pre-specified in the protocol, this study is not intended to be analyzed by arm for most analyses and data collection. Analysis for all arms will be combined for overall survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 21
months | 7.2 [4.4 to 13.7]

11. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS will summarized using the Kaplan-Meier method.
Time Frame: Up to 4 years
Population: As pre-specified in the protocol, this study is not intended to be analyzed by arm for most analyses and data collection. Analysis for all arms will be combined for progression free survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 21
months | 3.0 [1.8 to 4.9]

12. Secondary Outcome: Change in Component Phenolic Levels in Urine
Description: as for outcome 4
Time Frame: Baseline to up to 8 weeks
Measure: Mean (Standard Error); unit: ug/ml
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 20
ug/ml
  Baseline | 0.4 (7.9)
  Week 4 | 19.7 (8.2)
  Week 8 | 16.6 (8.6)

13. Secondary Outcome: Change in Component Phenolic Levels in Blood
Description: as for outcome 4
Time Frame: Baseline to up to 8 weeks
Population: Outcome measure was not measured
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 0

14. Secondary Outcome: Change in Quality of Life and Fatigue in Cancer Patients Taking MGE as Measured by PROMIS-Fatigue SF
Description: A mixed model ANOVA model will be fit with phenolic level as the outcome and time (baseline, every 4 weeks) as a fixed effect and subject as a random effect. Contrasts will be use to estimate changes from baseline to each follow-up time period. A 6-item questionnaire with T-score responses ranging from a minimum of 33.4 to a maximum of 76.8. Higher scores equals more of the concept being measured.
Time Frame: Baseline to up to 1 year
Population: As pre-specified in the protocol, this study is not intended to be analyzed by arm for most analyses and data collection. Analysis for all arms will be combined for change in quality of life. Not all participants completed intervention at the week 4 and week 8 time frames to be analyzed
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 21
T-score
  Baseline | 56.2 (2.5)
  Week 4: number analyzed (Participants) | 19
  Week 4 | 57.3 (2.6)
  Week 8: number analyzed (Participants) | 13
  Week 8 | 55.3 (2.7)
Statistical Analysis 1: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Test type: Other; p = 0.67, ANOVA

15. Secondary Outcome: Change in Systemic Cytokine Levels (Log IL-8)
Description: as for outcome 7
Time Frame: Baseline to up to 8 weeks
Population: Arms were combined for cytokine and phenolic analyses as pre-specified per protocol
Measure: Least Squares Mean (Standard Error); unit: log pg/mL
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 19
log pg/mL
  Baseline Log IL-8 | 1.49 (0.16)
  Week 4 Log IL-8 | 1.32 (0.17)
  Week 8 Log IL-8 | 1.40 (0.17)
Statistical Analysis 1: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Baseline v. 4 weeks log IL-8; Test type: Other; p = 0.119, ANOVA
Statistical Analysis 2: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Baseline v. 8 weeks log IL-8; Test type: Other; p = 0.414, ANOVA

16. Secondary Outcome: Change in Systemic Cytokine Levels (Log VEGF)
Description: as for outcome 7
Time Frame: Baseline to up to 8 weeks
Population: Arms were combined for cytokine and phenolic analyses as pre-specified per protocol
Measure: Least Squares Mean (Standard Error); unit: log pg/mL
Arm/Group | Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS
Number analyzed (Participants) | 19
log pg/mL
  Baseline Log VEGF | 2.78 (0.23)
  Week 4 Log VEGF | 2.81 (0.23)
  Week 8 Log VEGF | 2.84 (0.23)
Statistical Analysis 1: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Baseline v. 4 weeks p value log VEGF; Test type: Other; p = 0.851, ANOVA
Statistical Analysis 2: Comparison: Treatment (Muscadine Grape Skin Extract) FOR ALL ARMS; Baseline vs. 8 weeks p value log VEGF; Test type: Other; p = 0.688, ANOVA

ADVERSE EVENTS:
Time Frame: One year
Groups:
- Arm 3 (Muscadine Grape Skin Extract) 3 Pills Times a Day; Arm 4 (Muscadine Grape Skin Extract) 4 Pills Times a Day; Arm 5 (Muscadine Grape Skin Extract) 5 Pills Times a Day: Patients receive muscadine grape skin extract PO BID. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing benefit from muscadine grape skin extract may continue treatment in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Muscadine Grape Skin Extract: Given PO
Arm/Group | Arm 1 (Muscadine Grape Skin Extract) 1 Pill Times a Day | Arm 2 (Muscadine Grape Skin Extract) 2 Pills Times a Day | Arm 3 (Muscadine Grape Skin Extract) 3 Pills Times a Day | Arm 4 (Muscadine Grape Skin Extract) 4 Pills Times a Day | Arm 5 (Muscadine Grape Skin Extract) 5 Pills Times a Day
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/6 | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 0/3 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Muscadine Grape Skin Extract) 1 Pill Times a Day (N=3) | Arm 2 (Muscadine Grape Skin Extract) 2 Pills Times a Day (N=6) | Arm 3 (Muscadine Grape Skin Extract) 3 Pills Times a Day (N=3) | Arm 4 (Muscadine Grape Skin Extract) 4 Pills Times a Day (N=3) | Arm 5 (Muscadine Grape Skin Extract) 5 Pills Times a Day (N=6)
Sudden death, not otherwise specified (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Only 21 participants were evaluable for adverse events during this reporting cycle. Additional adverse events will be included at end of study.
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Muscadine Grape Skin Extract) 1 Pill Times a Day (N=3) | Arm 2 (Muscadine Grape Skin Extract) 2 Pills Times a Day (N=6) | Arm 3 (Muscadine Grape Skin Extract) 3 Pills Times a Day (N=3) | Arm 4 (Muscadine Grape Skin Extract) 4 Pills Times a Day (N=3) | Arm 5 (Muscadine Grape Skin Extract) 5 Pills Times a Day (N=6)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 5 (5) — Only 21 participants were evaluable for adverse events during this reporting cycle. Additional adverse events will be included at end of study.
Eye disorders (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema, face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema, limbs (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions, other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue, other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusions (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT02583269/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT02583269/ICF_001.pdf